CLINICAL TRIAL: NCT02620371
Title: Efficacy and Safety of Ketamine Added to Local Anesthetic in Modified Pectoral Block for Management of Postoperative Pain in Patients Undergoing Modified Radical Mastectomy
Brief Title: Efficacy of Ketamine Added to Local Anesthetic in Modified Pectoral Block for Management of Postoperative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 226
Record Dates: First submitted 2015-11-27; First posted 2015-12-03 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (bupivacaine) (Placebo Comparator): 30 patients were given preoperative ultrasound guided, modified pectoral block (pecs II block) with local anesthetic(0.25% bupivacaine)
  Interventions: Procedure: modified pectoral block
- (bupivacaine, ketamine) (Active Comparator): 30 patients were given preoperative ultrasound guided, modified pectoral block (pecs II block) with local anesthetic(0.25% bupivacaine plus ketamine 1 mg/kg) .
  Interventions: Procedure: modified pectoral block

INTERVENTIONS:
Procedure: modified pectoral block — Modified Pecs block was performed under general anesthesia, and 15 min. before skin incision. We performed the modified Pecs block or the " Pecs II block" by using a two needle approach instead of one. The first puncture is a Pecs I block with 10 ml of local anesthetic injected between the two pectoralis muscles, and the second puncture injects 20 ml of local anesthetic between the Pectoralis minor muscle and the serratus muscle. This breaks through the 'axillary door' and will reach the long thoracic nerve and reliably at least two intercostal nerves.
  We used A high frequency linear US probe is used for this block. a broadband linear array probe, with an imaging depth of 3-4cm. starting from the lateral third of the clavicle and moving distally and laterally to the mid axillary line.
  Other Names: pecs II block

SUMMARY:
This study aims to compare the analgesic efficacy and safety of local bupivacaine alone versus bupivacaine plus ketamine in ultrasound guided modified Pecs block in patients undergoing breast cancer surgery.

DETAILED DESCRIPTION:
This randomized Clinical trial was approved by the ethics committee of South Egypt Cancer Institute, Assuit University, Assuit, Egypt. Sixty patients aged 18 - 60 years, American Society of Anesthesiologists (ASA) class I-II, with body weight of 50 - 90 kg and arranged for modified radical mastectomy) were enrolled in this study. Patients with a history of bleeding diathesis, relevant drug allergy, opioid dependence, morbid obesity, sepsis, prior surgery in the supraclavicular, infraclavicular or axillary regions, alcohol or drug abuse and those with psychiatric illnesses that would interfere with perception and assessment of pain were excluded from the study.

Preoperatively, patients were taught how to evaluate their own pain intensity using the Visual Analog Scale (VAS), scored from 0-10 (where 0= no pain and 10=worst pain imaginable), and whenever (during the follow up period) VAS points to a value ≥ 3. Analgesia comprised PCA with an initial morphine bolus of 0.1mg/kg once pain expressed by the patient or if VAS ≥ 3 followed by 1mg boluses with a lockout period a 5 minute. The time to first request for analgesia and the total analgesic consumption in the first 24 hours were recorded.

On arrival to the operating room, an intravenous line was inserted. Monitoring included electrocardiography (ECG), non-invasive blood pressure (NIBP), arterial oxygen saturation (Sao2) and end-tidal carbon- dioxide were applied.

Anesthesia was induced for all participating patients with 2 μg/kg fentanyl, 2-3 mg/kg propofol and 1.5 mg/kg lidocaine. Endotracheal intubation was facilitated by 0.15 mg/kg cis-atracurium. Anesthesia was maintained by 1-1.5 MAC isoflurane in 50% oxygen / air mixture and 0.03 mg/kg cisatrcurium respectively in ventilation parameters to maintain on ETco2 of approximately 35- 40 mmHg. Ultrasound guided pecs block then performed

Patients were randomly assigned into 2 groups (using a randomization-computer program), 30 patients in each:

Group I (Bupivacaine group): patients were given ultrasound guided, modified Pecs block with 30 mL of 0.25% bupivacaine divided into 10 ml injected between the two pectoralis muscles on the interfascial plane, and 20 ml injected between the Pectoralis minor muscle and the serratus muscle.

Group II (Bupivacaine + ketamine group) : patients were given ultrasound guided, modified Pecs block with 30 ml of 0.25% bupivacaine plus ketamine (1 mg/kg) divided into 10 ml injected between the two pectoralis muscles on the interfascial plane , and 20 ml injected between the Pectoralis minor muscle and the serratus muscle.

Modified Pecs block was performed under general anesthesia, and 15 min. before skin incision. We performed the modified Pecs block or the " Pecs II block" by using a two needle approach instead of one. The first puncture is a Pecs I block with 10 ml of local anesthetic injected between the two pectoralis muscles, and the second puncture injects 20 ml of local anesthetic between the Pectoralis minor muscle and the serratus muscle. This breaks through the 'axillary door' and will reach the long thoracic nerve and reliably at least two intercostal nerves.

We used a broadband linear array probe, with an imaging depth of 3-4cm. starting from the lateral third of the clavicle and moving distally and laterally to the mid axillary line.

At the end of surgery, reversal of muscle relaxant was done using neostigmine (0.04 mg/kg) and atropine (0.01 mg/kg). After extubation; all patients were transmitted to post anesthesia care unit (PACU).

Each patient in both groups was followed up and assessed at baseline, 1h, 2h, 4h, 6h , 12h , 24h, 48h postoperatively for: Vital signs (The patients' heart rate, non invasive arterial blood pressure, respiratory rate and oxygen saturation), Post operative pain where the severity of pain was assessed using VAS score, the time to first request of rescue analgesia and total morphine consumption in the 48 hours.

Potential side effects, including, sedation by sedation score of 0-4 (0 = patient fully awake; 1 = patient somnolent and responsive to verbal commands; 2 = patient somnolent and responsive to tactile stimulation; and 3 = patient asleep and responsive to painful stimulation; 4 = not arousable), chest pain, nausea, vomiting (treated by IV boluses of metochlopromide 10 mg), and psychological complications (hallucination, delirium, dreams, nystagmus, dissociative effects) were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I-II
* Body weight of 50 - 90 kg

Exclusion Criteria:

* History of bleeding diathesis
* Relevant drug allergy, opioid dependence
* Morbid obesity, sepsis
* prior surgery in the supraclavicular, infraclavicular or axillary regions,
* Alcohol or drug abuse
* Those with psychiatric illnesses that would interfere with perception and assessment of pain

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | first 48 hours postoperatively
  Total morphine consumption in mg in the first 48 hours postoperatively

SECONDARY OUTCOMES:
first request of rescue analgesia | 48 hours postoperatively
  first request of analgesia in hours in the first 48 hrs postoperative
the severity of pain was assessed using VAS score | 48 hours postoperatively
  he severity of pain was assessed using VAS score in 48 hours postoperative

OTHER OUTCOMES:
Potential side effects | 48 hours postoperatively
  Potential side effects, including, sedation by sedation score of 0-4 (0 = patient fully awake; 1 = patient somnolent and responsive to verbal commands; 2 = patient somnolent and responsive to tactile stimulation; and 3 = patient asleep and responsive to painful stimulation; 4 = not arousable), chest pain, nausea, vomiting (treated by IV boluses of metochlopromide 10 mg), and psychological complications (hallucination, delirium, dreams, nystagmus, dissociative effects)

CONTACTS AND LOCATIONS:
Overall Officials: UNVERSITY, Principal Investigator — ASSUIT
Locations (1):
- South Egypt Cancer Instuite, Asyut, Egypt

REFERENCES:
- [Derived] Othman AH, El-Rahman AM, El Sherif F. Efficacy and Safety of Ketamine Added to Local Anesthetic in Modified Pectoral Block for Management of Postoperative Pain in Patients Undergoing Modified Radical Mastectomy. Pain Physician. 2016 Sep-Oct;19(7):485-94. PMID 27676665